CLINICAL TRIAL: NCT03310658
Title: Zip-Stitch™ for Vaginal Cuff Closure in Total Laparoscopic Hysterectomy: First in Human Ease of Use Study
Brief Title: Zip-Stitch™ for Vaginal Cuff Closure in Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZSX Medical LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ZHP01-1.0
Record Dates: First submitted 2017-09-26; First posted 2017-10-16 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2017-10

CONDITIONS: Total Laparoscopic Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Study Site: UANL (Experimental): As the only study arm, 10 enrolled subjects received vaginal cuff closure with the Zip-Stitch Soft Tissue Closure System as part of Total Laparoscopic Hysterectomy.
  Interventions: Device: Zip-Stitch Soft Tissue Closure System

INTERVENTIONS:
Device: Zip-Stitch Soft Tissue Closure System — The novel Zip-Stitch System employed a laparoscopic applicator, a series of bio-absorbable clips, and an application procedure to close the vaginal cuff during otherwise standard of care total laparoscopic hysterectomy.

SUMMARY:
ZSX Medical completed enrollment in its First in Human Ease of Use study in May of 2017, in Monterrey Mexico. The purpose of this study is to demonstrate the ease of use of Zip-Stitch™, to generate first in human data, and to refine surgical technique of the device.

Ten subjects were enrolled and received total laparoscopic hysterectomies, including vaginal cuff closure with the Zip-Stitch™ system during their otherwise standard care. Procedures took place over the course of one week. Subjects had in person follow-up appointments at 1 and 6 weeks. Subjects are continuing follow-up through a one-year extension period which will end in May 2018.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated Informed Consent Form
* Stated willingness to comply with all study procedures, including participation in follow-up visits and telephonic follow-up
* Female, age 18 years or older
* Indicated for Total Laparoscopic Hysterectomy

Exclusion Criteria:

* HIV
* Hepatitis C
* Diabetics
* Use of systemic corticosteroids
* History of pelvic irradiation
* Active infection
* History of bleeding problems/hemophilia
* Cancer
* Cases in which vaginal cuff closure is intended to be performed robotically
* Pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Device Ease of Use | Immediately following procedure
  Ease of Use of the Zip-Stitch Soft Tissue Closure System during Total Laparoscopic Hysterectomy. Assessed following surgery by standardized surgeon interview.

SECONDARY OUTCOMES:
Vaginal Cuff Closure | During procedure.
  Assessment of quality of vaginal cuff closure following uterine excision. Performed by surgeon as operative standard of care.
Vaginal Cuff Closure Time | During Procedure.
  Procedural time from uterine excision to successful vaginal cuff closure.
Total Surgical Time | During Procedure.
  Total procedural time.
Device Use Learning Curve assessed with a Surgeon Survey | Assessed immediately following study completion during surgeon survey.
  Investigation of change in effectiveness of device implementation as assessed by change in efficiency of device use.
Sexual Discomfort | Assessed at 1 and 6 week follow-up visits.
  Measurement of subject discomfort during sexual activity following completion of surgical procedure. Assessed with 1-10 scale (1 = No Pain, 10 = Most Pain).

CONTACTS AND LOCATIONS:
Overall Officials: Dan Mazzucco, PhD, Study Director — ZSX Medical LLC
Locations (1):
- Hospital Universitario: Universidad Autónoma de Nuevo León de Monterrey, Monterrey, Nuevo León, Mexico